CLINICAL TRIAL: NCT00986206
Title: Development of an Assay for the Early Detection of Ovarian Cancer.
Brief Title: Lysophosphatidic Acid Assay in Patients With Ovarian Cancer or Who Are at Risk for Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Richard G. Moore, MD, Gynecologic Oncologist, Women and Infants Hospital of Rhode Island
Other Study IDs: WIHRI-09-0030; CDR0000655148 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-09-26; First posted 2009-09-29 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Ovarian Cancer
Keywords: ovarian epithelial cancer; BRCA1 mutation carrier; BRCA2 mutation carrier; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker testing: Collect serum for biomarker testing for LAP and HE4 and discovery of new biomarkers.
  Interventions: Diagnostic Test: Biomarker LPA and HE4

INTERVENTIONS:
Diagnostic Test: Biomarker LPA and HE4 — Non Interventional Trial

SUMMARY:
RATIONALE: Screening tests, such as the lysophosphatidic acid assay, may help doctors find cancer cells early and plan better treatment for ovarian cancer.

PURPOSE: This clinical trial is studying using the lysophosphatidic acid assay to see how well it works in early detection of ovarian cancer in patients with ovarian cancer or who are at risk for ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To validate a new assay for lysophosphatidic acid (LPA) in early detection of ovarian cancer.

Secondary

* To estimate the risk of finding ovarian cancer at the time of surgery in pre- and post-menopausal women presenting with a pelvic mass and compare LPA results from both surgical patient groups with those from "normal", disease-free women at high-risk of ovarian cancer.

Tertiary

* To examine the response to primary adjuvant treatment and recurrence of disease.
* To evaluate urine levels of CA125 and LPA to determine their ability to estimate the risk of cancer at the time of surgery in patients presenting with a pelvic mass. (exploratory)

OUTLINE: Blood and urine samples are collected before or on the day of surgery; before, during, and after completing chemotherapy; or at a clinic visit. Samples are tested for concentrations of CA125 and lysophosphatidic acid (LPA) using a new assay and compared to liquid chromatography/electrospray ionization-tandem mass spectrometry results. Remaining serum, plasma, and urine is stored frozen for future research evaluation of other novel biomarkers for the diagnosis and prognosis of cancer.

After completion of study, patients are followed up periodically for approximately 5 years.

PROJECTED ACCRUAL: A total of 500 surgical patients, 100 cancer patients undergoing first-line therapy, and 40 disease-free women who are known BRCA-mutation carriers will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Presenting to a gynecological oncologist with a unilateral or bilateral pelvic mass (defined as a simple, complex, or a solid ovarian/pelvic mass) and scheduled to undergo surgery
  * Newly diagnosed epithelial ovarian cancer and undergoing first-line chemotherapy
  * History of epithelial ovarian carcinoma status post-primary chemotherapy treatment, currently in clinical remission according to the following criteria:

    * Absence of symptoms that may be related to disease
    * Imaging without abnormalities ≥ 1 cm suspicious for disease (no ascites)
    * CA125 obtained twice at least 3 weeks apart and not increasing by 50% and < 40 units/mL
  * Known BRCA mutations and intact ovaries (no prior bilateral salpingo-oophorectomy)
* No synchronous primary endometrial cancer or a past history of primary endometrial cancer, unless all of the following conditions are met:

  * Stage not greater than IB
  * No more than superficial myometrial invasion, without vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesions
* No epithelial ovarian carcinoma of low malignant potential (borderline carcinomas)
* Patients of any stage who have recurred and are in second chemotherapy induced remission are not eligible

PATIENT CHARACTERISTICS:

* Pre- or post-menopausal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancies within the past 5 years, with the exception of nonmelanoma skin cancer
* No septicemia, severe infection, or acute hepatitis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to any portion of the abdominal cavity or pelvis
* No prior chemotherapy for another malignancy

Inclusion Criteria:

* Eligible Patients
* Patients age ≥ 21 years
* Patients with a diagnosis of a pelvic mass (defined as a simple, complex or a solid ovarian / pelvic mass) who are scheduled to undergo surgery.
* Patients with a new diagnosis of epithelial ovarian carcinoma undergoing primary chemotherapy treatment.
* Patients with a history of epithelial ovarian carcinoma status post primary chemotherapy treatment, currently in clinical remission.
* Patients with a known BRCA mutation and who have NOT undergone a bilateral salpingo-oophorectomy.
* Clinical remission should require all of following:
* Absence of symptoms that may be related to disease;
* Imaging without abnormalities greater then or equal to 1 cm suspicious for disease (no ascites);
* CA 125 obtained x 2 at least 3 weeks apart and not increasing by 50% and < 40 units/mL.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Women of childbearing potential must have a negative pregnancy test. They as well as their partners must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.

Exclusion Criteria:

* Ineligible Patients
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients with synchronous primary endometrial cancer or a past history of primary endometrial cancer are excluded, unless all of the following conditions are met: Stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO Grade 3 lesions.
* Patients with epithelial ovarian carcinoma of low malignant potential (Borderline carcinomas).
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis or have received chemotherapy for another malignancy.
* Patients of any stage who have recurred and are in second chemotherapy induced remission.
* Patients with septicemia, severe infection, or acute hepatitis.
* Patients who are pregnant or lactating.

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women presenting with a pelvic mass and scheduled to undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2009-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Validation of a new assay for lysophosphatidic acid (LPA) | 5 years
  To develop a serum or plasma based assay to quantitate LPA levels

SECONDARY OUTCOMES:
Risk of finding ovarian cancer at the time of surgery in pre- and post-menopausal women | 5 years
  To evaluate a quantitative serum LPA assay and correlate serum LPA levels in pre and post menopausal women with benign and malignant ovarian tumors.
LPA results in pre- and post-menopausal women and women at high-risk of ovarian cancer | 5 years
  To measure serum LPA levels in pre and postmenopausal women

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Moore, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States